CLINICAL TRIAL: NCT05688397
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluate the Vaginal Colonization Capacity, Safety, and Tolerability of Two New Strains of L. Gasseri and L. Crispatus When Administered Orally in Healthy Female Volunteers
Brief Title: Evaluation of the Vaginal Colonization of Two New Lactobacillus Strains After Oral Administration in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: OLIVIA
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: probiotics
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1 (Experimental): L. gasseri oral capsule
  Interventions: Dietary Supplement: Experimental 1
- Experimental 2 (Experimental): L. gasseri + L. crispatus oral capsule
  Interventions: Dietary Supplement: Experimental 2
- Placebo (Placebo Comparator): Maltodextrin (E1400, qs) oral capsule once a day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Experimental 1 — L. gasseri oral capsule once a day (1 x 10^9 CFU/day) for 18 days starting the next day after menstruation is over
  Other Names: Probiotic
  Arms: Experimental 1
Dietary Supplement: Experimental 2 — L. gasseri and L. crispatus oral capsule once a day (1.5 x 10^9 CFU/day) for 18 days starting the next day after menstruation is over
  Other Names: Probiotic mixture
  Arms: Experimental 2
Dietary Supplement: Placebo — One maltodextrin-containing capsule a day for 18 days starting the next day after menstruation is over
  Arms: Placebo

SUMMARY:
Randomized study to determine whether the vaginally isolated strains of Lactobacillus gasseri and/or Lactobacillus crispatus can colonize the vagina when taken orally for 18 days. Secondary outcomes comprise evaluation of safety, tolerability, impact on vaginal microbiota and vaginal pH

DETAILED DESCRIPTION:
Double blind, randomized, placebo-controlled biomedical research study to determine whether supplementation with the vaginally isolated strains of Lactobacillus gasseri and/or Lactobacillus crispatus can colonize the vagina. Healthy women who meet inclusion and exclusion criteria will be randomized 1.5:1.5:1 to one of the following study groups: group one will receive L.gasseri for 18 days (1 capsule/day), group two will recieve the combination of L.gasseri and L.Crispatus for 18 days (1 capsule/day) and the other will receive placebo, starting the day after menstruation is over. Main study outcome will be colonization throughout the study, which will be determined by analysis of specific strains by qPCR. Secondary outcomes comprise comprise evaluation of tolerability, impact on vaginal microbiota, vaginal pH and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Reproductive age 18-45 years

Exclusion Criteria:

* Vaginal infection or symptoms (AMSEL criteria).
* Relevant disease (immunodeficiency, cervicovaginal pathology, diabetes, estrogen-dependent tumors, inflammatory bowel disease, atrophic vaginitis, pancreatitis)
* Suffer from chronic diarrhea or constipation or short bowel syndrome,
* Having taken systemic or vaginal antibiotics or antifungals during the month prior to study entry.
* Pregnant women or willing to be during the study, lactating women.
* Having taken another probiotic during the month prior to study entry orally or vaginally. This includes food supplements or foods supplemented with probiotics such as Actimel, Activia or similar.
* Intake of immunomodulators or systemic corticosteroids.
* History of alcohol or drug abuse.
* Menopausal women.
* Use of the IUD.
* Use of spermicides or vaginal lubricants during the month prior to study entry.
* Very irregular periods or low probability of going at least 18 days without menstruation (short cycles).
* Have participated in a clinical trial during the month prior to entering the study.
* Not being able to follow or understand study procedures. This includes not being willing to maintain sexual abstinence during the 24 hours prior to each vaginal sample collection.
* Any other condition not compatible with the study according to the investigators

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Colonization of L. crispatus strain in the vagina | 0,15 or 18 days
  Change in the concentration of L. crispatus strain throughout study period measured by qPCR in samples obtained with vaginal swab
Colonization of L. gasseri strain in the vagina | 0,15 or 18 days
  Change in the concentration of L. gasseri strain throughout study period measured by qPCR in samples obtained with vaginal swab

SECONDARY OUTCOMES:
Vaginal colonization of L. gasseri strain | Day 0, 3, 6, 9, 12, 15
  Change in the vaginal concentration of L. gasseri strain measured by qPCR versus baseline
Vaginal colonization of L. crispatus strain | Day 0, 3, 6, 9, 12, 15
  Change in the vaginal concentration of L. crispatus strain measured by qPCR versus baseline
Vaginal microbiota composition | Day 0, 6, 12 and 15 or 18
  Change in vaginal microbiota composition measured by 16S rRNA sequencing analysis in samples obtained from vaginal swabs
Perianal concentration of L. crispatus strain | Day 0, 9 and 15 or 18
  Change in the perianal concentration of L. crispatus strain measured by qPCR
Perianal concentration of L. gasseri strain | Day 0, 9 and 15 or 18
  Change in the perianal concentration of L. gasseri strain measured by qPCR
Vaginal pH | Day 0, 3, 6, 9, 12, 15, 18
  Change in vaginal pH throughout study period measured by pH test strip
Gastrointestinal symptoms | day 0, day 18
  Gastrointestinal manifestations measured on a 4-point scale: 0 = none , 1 = mild, 2 = moderate, and 3 = severe.
Adverse events | 18 days
  Frequency of adverse events throughout study period
Satisfaction with the product | Day 18
  Evaluation of the satisfaction with the product through the Treatment Satisfaction Questionnaire for Medication (TSQM)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Maria Aldea Perona, PhD, Principal Investigator — Instituto Hospital del Mar de Investigaciones Médicas
Locations (1):
- Instituto Hospital del Mar de Investigaciones Médicas, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez M, Armengol E, Del Casale A, Campedelli I, Aldea-Perona A, Perez Otero M, Rodriguez-Palmero M, Espadaler-Mazo J, Huedo P. Lactobacillus gasseri CECT 30648 shows probiotic characteristics and colonizes the vagina of healthy women after oral administration. Microbiol Spectr. 2025 Sep 2;13(9):e0021125. doi: 10.1128/spectrum.00211-25. Epub 2025 Aug 7. PMID 40772934